CLINICAL TRIAL: NCT04014244
Title: Efficacy of Dextrose Injections, Corticosteroids Injections and Surgical Release for Treatment of the Carpal Tunnel Syndrome: a Prospective, Randomized, Double-blind Controlled Trial
Brief Title: Dextrose, Corticosteroids and Surgical Release in Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Gregor Omejec, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Treatment SZP
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Nervous System Diseases; Nerve Compression Syndromes; Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Electromyography; Ultrasonography; Surgery; Dextrose; Corticosteroids
MeSH Terms: conditions — Peripheral Nervous System Diseases; Nerve Compression Syndromes; Carpal Tunnel Syndrome | interventions — Glucose; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Patients with bilateral CTS symptoms and EDx mild to moderate CTS will be included. In the first part of the study examiner will randomize substance for left hand infiltration using a dice (odd number - corticosteroids; even number - 5% glucose). Right hand will be infiltrated with the remaining substance. In the second part of the study examiner will randomize treatment procedure for left hand using a dice (odd number - corticosteroids or 5% glucose; even number - surgery). Substance for injection will be determined according to the results of the first part of the study - more effective one, or in case of non-inferiority 5% glucose will be used. In all patients included in the second part of the study surgical release will be performed by the same plastic surgeon. Both treatments will be performed maximally 2 months after diagnosis, with maximum period between them of 1 week.
Who Masked: Participant, Investigator
Masking Description: Each of three investigators performing one part of diagnostic evaluation (history and focal neurologic examination, EDx and (3) ultrasonographic (US) studies) will be blinded for findings of other parts of evaluation. Furthermore, patients will be blinded for laterality of the injected substance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroids vs. Dextrose (Experimental): In the first part of the study examiner will randomize substance for left hand infiltration using a dice (odd number - corticosteroids; even number - 5% glucose). Right hand will be infiltrated with the remaining substance.
  Interventions: Drug: Corticosteroid vs. Dextrose
- Corticosteroids or Dextrose vs. Surgery (Experimental): In the second part of the study examiner will randomize treatment procedure for left hand using a dice (odd number - corticosteroids or 5% glucose; even number - surgery). Substance for injection will be determined according to the results of the first part of the study - more effective one, or in case of non-inferiority 5% glucose will be used. Surgical release will be performed by the same plastic surgeon. Both treatments will be performed maximally 2 months after diagnosis, with maximum period between them of 1 week.
  Interventions: Procedure: Corticosteroid or Dextrose vs. Surgery

INTERVENTIONS:
Drug: Corticosteroid vs. Dextrose — US guided injection of corticosteroid in one hand and 5% glucose in the other will be performed in accordance with randomization. In a syringe both substances will be diluted using 0.9% NaCl to a total injection volume of 6 ml. In-plane ulnar approach will be used to visualize the median nerve at the level of the pisiform bone. A standard 23 gauge needle will be inserted in the carpal tunnel with the needle tip positioned between retinaculum and median nerve.
  Other Names: Triamcinolone injections versus 5% dextrose
  Arms: Corticosteroids vs. Dextrose
Procedure: Corticosteroid or Dextrose vs. Surgery — Injection will be performed unilaterally, after randomization of sides, by the same examiner as in the first part of the study. In all patients included in the second part of the study surgical release will be performed by the same plastic surgeon. The procedure will be performed under local anesthesia, following the same standard protocol. Both treatments will be performed maximally 2 months after diagnosis, with maximum period between them of 1 week.
  Other Names: Triamcinolone injections or 5% dextrose versus Carpal tunnel release
  Arms: Corticosteroids or Dextrose vs. Surgery

SUMMARY:
The objective of the present study is to compare the effectiveness of 5% dextrose, local corticosteroids injections and surgical release in patients with electrodiagnostically (EDx) mild to moderate carpal tunnel syndrome (CTS). The investigators hypothesize that in patients with mild to moderate CTS (1) local 5% dextrose injections is non-inferior to local corticosteroid injections at 12 months after treatment, and that (2) local 5% dextrose injections are of non-inferior effectiveness compared to surgical release at 6 months.

DETAILED DESCRIPTION:
Surgical release of the carpal ligament is a standard treatment of the median nerve entrapment at the wrist. Local corticosteroid injections are also an established alternative, particularly for EDx mild or moderate CTS, although majority of patients still needs surgical decompression within 1 year. Majority of studies concluded that after more than 6 months of treatment surgical decompression is better than local corticosteroids injections. Furthermore, corticosteroids also have a number of side effects, including crystal induced synovitis, tendon rupture, axon and myelin degeneration, soft tissue atrophy, skin thinning, steroid flare and hot flushes. Therefore, it would be very useful to have an effective alternative substance for injections, without these problems. Perineural injection of dextrose also seems to be a promising treatment for entrapment neuropathies. To date only two studies investigated the effectiveness of 5% dextrose injections in patients with CTS. Authors concluded that this is an effective treatment, that is for patients with mild or moderate CTS even more beneficial than corticosteroid injections at 6 months follow-up. It was suggested that perineural injection of 5% dextrose decreases neurogenic inflammation. As 5% dextrose has osmolarity similar to normal saline, this formulation seems particularly promising. These expectations were supported in studies including animals and humans reporting no harmful effects.

ELIGIBILITY:
Inclusion Criteria (subject diagnosed as CTS if meeting criterion 1 + at least one of criteria 2 or 3):

1. numbness and tingling in at least two out of the first four digits;
2. symptoms exacerbated during the night or in the morning, on holding the objects or repetitive use of the hand;
3. symptoms relieved by shaking the hand or reposition of the arm.

In addition to these clinical criteria for recruitment EDx confirmation will also be needed. Only patients with bilateral EDx mild to moderate CTS will be included.

Exclusion Criteria:

1. polyneuropathy, symptoms of polyneuropathy, and all conditions causing polyneuropathy (e.g., diabetes);
2. multiple mononeuropathy (e.g., hereditary neuropathy with liability to pressure palsies, syndrome Lewis Sumner);
3. motor neuron disorders (e.g., monomelic amyotrophy, amyotrophic lateral sclerosis - ALS);
4. brachial plexopathy;
5. other focal neuropathies affecting upper limbs (e.g., other median neuropathies, ulnar neuropathies, thoracic outlet syndrome); or
6. previous surgery or local injections for CTS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Score | 1 years
  The Visual Analog Scale (VAS) will be used to assess severity of digital paresthesia/dysesthesia and wrist or hand pain on 11-point grading scale. Scores ranges from from 0 to 10 points, with higher scores indicating greater severity of CTS symptoms (0 - no symptoms; 10 - extremely severe symptoms).

SECONDARY OUTCOMES:
Global Assessment of Treatment Results | 1 years
  At 1-, 3-, 6- and 12-month follow-up assessments, CTS symptoms relief after treatment will be evaluated and categorized as one of the following: (1) much improved, (2) improved, (3) no change, (4) worse, or (5) much worse. Patients in category 1 or 2 will be considered to have effective treatment.
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) Score | 1 years
  The self-administered Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) (Levine et al., 1993) includes 2 subscales of symptoms severity (11 questions) and functional status (8 questions). It is the most commonly used measurement for CTS. Scores ranges from 0 to 5 points for each question, with higher scores indicating greater severity and dysfunction.
Median Nerve Distal Motor Latency (DML) | 1 years
  Distal motor latency (DML) will be measured with median nerve stimulation 8 cm proximal to the active electrode over the abductor pollicis brevis muscle in each hand before and at 1-, 3, 6 and 12 months after treatment.
Ulnar and Median Antidromic Sensory Nerve Action Potentials (SNAPs) | 1 years
  Ulnar and median antidromic sensory nerve action potentials (SNAPs) from 4th finger will be recorded on the nerve stimulation 14 cm proximal to recording electrode placed at the middle of the first phalange and SNAP latency difference calculated.
Median Nerve Cross-sectional Area (CSA) | 1 years
  Cross-sectional Area (CSA) of the median nerve will be measured at the wrist and 15 cm proximal at the forearm using a trace method with exclusion of the hyperechoic rim.
Palmar Bowing of the Flexor Retinaculum | 1 years
  Palmar bowing of the flexor retinaculum is a measure used to quantify the internal pressure exerted on the retinaculum from the contents within the carpal tunnel as the perpendicular distance between flexor retinaculum and tangential line between the tip of the pisiform and scaphoid bone.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Department of Neurology, Institute of Clinical Neurophysiology, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verdugo RJ, Salinas RS, Castillo J, Cea JG. Surgical versus non-surgical treatment for carpal tunnel syndrome. Cochrane Database Syst Rev. 2003;(3):CD001552. doi: 10.1002/14651858.CD001552. PMID 12917909
- [Background] Marshall S, Tardif G, Ashworth N. Local corticosteroid injection for carpal tunnel syndrome. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD001554. doi: 10.1002/14651858.CD001554.pub2. PMID 17443508
- [Background] Atroshi I, Flondell M, Hofer M, Ranstam J. Methylprednisolone injections for the carpal tunnel syndrome: a randomized, placebo-controlled trial. Ann Intern Med. 2013 Sep 3;159(5):309-17. doi: 10.7326/0003-4819-159-5-201309030-00004. PMID 24026316
- [Background] Andreu JL, Ly-Pen D, Millan I, de Blas G, Sanchez-Olaso A. Local injection versus surgery in carpal tunnel syndrome: neurophysiologic outcomes of a randomized clinical trial. Clin Neurophysiol. 2014 Jul;125(7):1479-84. doi: 10.1016/j.clinph.2013.11.010. Epub 2013 Nov 23. PMID 24321619
- [Background] Ly-Pen D, Andreu JL, de Blas G, Sanchez-Olaso A, Millan I. Surgical decompression versus local steroid injection in carpal tunnel syndrome: a one-year, prospective, randomized, open, controlled clinical trial. Arthritis Rheum. 2005 Feb;52(2):612-9. doi: 10.1002/art.20767. PMID 15692981
- [Background] Ly-Pen D, Andreu JL, Millan I, de Blas G, Sanchez-Olaso A. Comparison of surgical decompression and local steroid injection in the treatment of carpal tunnel syndrome: 2-year clinical results from a randomized trial. Rheumatology (Oxford). 2012 Aug;51(8):1447-54. doi: 10.1093/rheumatology/kes053. Epub 2012 Mar 30. PMID 22467087
- [Background] Celik G, Ilik MK. Effects of Two Different Treatment Techniques on the Recovery Parameters of Moderate Carpal Tunnel Syndrome: A Six-Month Follow-up Study. J Clin Neurophysiol. 2016 Apr;33(2):166-70. doi: 10.1097/WNP.0000000000000243. PMID 26657237
- [Background] Peters-Veluthamaningal C, Winters JC, Groenier KH, Meyboom-de Jong B. Randomised controlled trial of local corticosteroid injections for carpal tunnel syndrome in general practice. BMC Fam Pract. 2010 Jul 29;11:54. doi: 10.1186/1471-2296-11-54. PMID 20670438
- [Background] Ustun N, Tok F, Yagz AE, Kizil N, Korkmaz I, Karazincir S, Okuyucu E, Turhanoglu AD. Ultrasound-guided vs. blind steroid injections in carpal tunnel syndrome: A single-blind randomized prospective study. Am J Phys Med Rehabil. 2013 Nov;92(11):999-1004. doi: 10.1097/PHM.0b013e31829b4d72. PMID 23811617
- [Background] Lee JY, Park Y, Park KD, Lee JK, Lim OK. Effectiveness of ultrasound-guided carpal tunnel injection using in-plane ulnar approach: a prospective, randomized, single-blinded study. Medicine (Baltimore). 2014 Dec;93(29):e350. doi: 10.1097/MD.0000000000000350. PMID 25546691
- [Background] Makhlouf T, Emil NS, Sibbitt WL Jr, Fields RA, Bankhurst AD. Outcomes and cost-effectiveness of carpal tunnel injections using sonographic needle guidance. Clin Rheumatol. 2014 Jun;33(6):849-58. doi: 10.1007/s10067-013-2438-5. Epub 2013 Nov 26. PMID 24277115
- [Background] Wang JC, Liao KK, Lin KP, Chou CL, Yang TF, Huang YF, Wang KA, Chiu JW. Efficacy of Combined Ultrasound-Guided Steroid Injection and Splinting in Patients With Carpal Tunnel Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 May;98(5):947-956. doi: 10.1016/j.apmr.2017.01.018. Epub 2017 Feb 14. PMID 28209506
- [Background] Wang PH, Tsai CL, Lee JS, Wu KC, Cheng KI, Jou IM. Effects of topical corticosteroids on the sciatic nerve: an experimental study to adduce the safety in treating carpal tunnel syndrome. J Hand Surg Eur Vol. 2011 Mar;36(3):236-43. doi: 10.1177/1753193410390760. Epub 2011 Jan 31. PMID 21282223
- [Background] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Tsai CK, Chen LC. Six-month Efficacy of Perineural Dextrose for Carpal Tunnel Syndrome: A Prospective, Randomized, Double-Blind, Controlled Trial. Mayo Clin Proc. 2017 Aug;92(8):1179-1189. doi: 10.1016/j.mayocp.2017.05.025. PMID 28778254
- [Background] Wu YT, Ke MJ, Ho TY, Li TY, Shen YP, Chen LC. Randomized double-blinded clinical trial of 5% dextrose versus triamcinolone injection for carpal tunnel syndrome patients. Ann Neurol. 2018 Oct;84(4):601-610. doi: 10.1002/ana.25332. Epub 2018 Oct 4. PMID 30187524
- [Background] Hashimoto K, Sakura S, Bollen AW, Ciriales R, Drasner K. Comparative toxicity of glucose and lidocaine administered intrathecally in the rat. Reg Anesth Pain Med. 1998 Sep-Oct;23(5):444-50. doi: 10.1016/s1098-7339(98)90025-6. PMID 9773695
- [Background] Sakura S, Chan VW, Ciriales R, Drasner K. The addition of 7.5% glucose does not alter the neurotoxicity of 5% lidocaine administered intrathecally in the rat. Anesthesiology. 1995 Jan;82(1):236-40. doi: 10.1097/00000542-199501000-00028. PMID 7832306
- [Background] Tsui BCH, Kropelin B. The electrophysiological effect of dextrose 5% in water on single-shot peripheral nerve stimulation. Anesth Analg. 2005 Jun;100(6):1837-1839. doi: 10.1213/01.ANE.0000153020.84780.A5. PMID 15920223
- [Background] Dufour E, Donat N, Jaziri S, Kurdi O, Couturier C, Dreyfus JF, Fischler M. Ultrasound-guided perineural circumferential median nerve block with and without prior dextrose 5% hydrodissection: a prospective randomized double-blinded noninferiority trial. Anesth Analg. 2012 Sep;115(3):728-33. doi: 10.1213/ANE.0b013e31825fa37d. Epub 2012 Jun 28. PMID 22745114
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] Ng AWH, Griffith JF, Lee RKL, Tse WL, Wong CWY, Ho PC. Ultrasound carpal tunnel syndrome: additional criteria for diagnosis. Clin Radiol. 2018 Feb;73(2):214.e11-214.e18. doi: 10.1016/j.crad.2017.07.025. Epub 2017 Aug 30. PMID 28859853
- [Background] Lee YS, Choi E. Ultrasonographic changes after steroid injection in carpal tunnel syndrome. Skeletal Radiol. 2017 Nov;46(11):1521-1530. doi: 10.1007/s00256-017-2738-y. Epub 2017 Aug 2. PMID 28770310
- [Background] Gonzalez-Suarez CB, Fidel BC, Cabrera JTC, Dela Cruz FC, Gesmundo MVT, Regala CFG, Saratan R, Suarez CG, Grimmer K. Diagnostic Accuracy of Ultrasound Parameters in Carpal Tunnel Syndrome: Additional Criteria for Diagnosis. J Ultrasound Med. 2019 Nov;38(11):3043-3052. doi: 10.1002/jum.15012. Epub 2019 Apr 17. PMID 30993769
- [Background] Smith J, Wisniewski SJ, Finnoff JT, Payne JM. Sonographically guided carpal tunnel injections: the ulnar approach. J Ultrasound Med. 2008 Oct;27(10):1485-90. doi: 10.7863/jum.2008.27.10.1485. PMID 18809959
- [Background] Scholten RJ, Mink van der Molen A, Uitdehaag BM, Bouter LM, de Vet HC. Surgical treatment options for carpal tunnel syndrome. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD003905. doi: 10.1002/14651858.CD003905.pub3. PMID 17943805